CLINICAL TRIAL: NCT02888275
Title: The Renal Protective Effect of the Dexmedetomidine in Pediatric Patients Undergoing Cardiac Surgery
Brief Title: Dexmedetomidine in Pediatric Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H1608-052-784
Record Dates: First submitted 2016-08-30; First posted 2016-09-05 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- DEX (Experimental): dexmedetomidine 1mcg/kg for 10min. loading and continuous infusion during the surgery 0.5mcg/kg/hr.
  Interventions: Drug: Dexmedetomidine
- no_DEX (Active Comparator): Normal saline 1mcg/kg for 10min. and continuous infusion during the surgery 0.5mcg/kg/hr.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Dexmedetomidine
  Arms: DEX
Drug: normal saline
  Arms: no_DEX

SUMMARY:
Dexmedetomidine is a selective α-2 receptor agonist with a sedative and cardiopulmonary profile that makes it an attractive anesthetic for pediatric patients with congenital heart disease (CHD). The aim of this study was to investigate the renal protective effect of dexmedetomidine in the perioperative setting in children with heart disease.

Total 144 pediatric patients allocated dexmedetomidine (DEX) and did not receive the drug (NoDEX) group.

The primary objective of this study was to assess the relationship between the use of intraoperative dexmedetomidine and the incidence of acute kidney injury in pediatric patients undergoing cardiopulmonary bypass. The secondary objective was to determine whether there was an association between dexmedetomidine use and duration of mechanical ventilation or cardiovascular ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing congenital cardiac surgery

Exclusion Criteria:

* history of allergy or anaphylaxis to study drug
* preexisting renal dysfunction (preoperative creatinine >1.5mg/dl)
* diabetes
* liver profile abnormality

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
serum creatinine | immediate after surgery, until discharge from the ICU, assessed up to 1 week.
  daily check the laboratory parameter.

SECONDARY OUTCOMES:
glomerular filtration rate | immediate after surgery, until discharge from the ICU, assessed up to 1 week.
  daily check the laboratory parameter.
Urine output | immediate after surgery, until discharge from the ICU, assessed up to 1 week.
  daily check the laboratory parameter.

CONTACTS AND LOCATIONS:
Locations (1):
- Jin-Tae Kim, Seoul, South Korea